CLINICAL TRIAL: NCT06770452
Title: A Single-arm Phase II Study of HRS-4642 With Nimotuzumab and Chemotherapy for First-line Treatment of Advanced Pancreatic Cancer Patients With KRAS G12D Mutations
Brief Title: HRS-4642 With Nimotuzumab and Chemotherapy for First-line Treatment of Advanced Pancreatic Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPT04
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Eligible patients will receive HRS-4642, combined with Nimotuzumab and AG regimen, predose regimen: HRS-4642 500mg intravenous infusion, D1,1200mg IV infusion, D8, every 3 weeks; Nimotuzumab 400mg intravenous infusion, D1,8, every 3 weeks; Albumin paclitaxel 125mg/m2 intravenous infusion, gemcitabine 1000mg / m2, D1,8, a cycle every 3 weeks until disease progression or toxicity intolerance.
  Interventions: Drug: HRS-4642; Drug: Nimotuzumab; Drug: gemcitabine + nab-paclitaxel

INTERVENTIONS:
Drug: HRS-4642 — HRS-4642 is a KRAS G12D inhibitor
Drug: Nimotuzumab — Nimotuzumab is a humanized IgG 1 monoclonal antibody targeting EGFR
Drug: gemcitabine + nab-paclitaxel — Albumin paclitaxel 125mg/m2 intravenous infusion, gemcitabine 1000mg / m2, D1,8, a cycle every 3 weeks

SUMMARY:
This study is a single-arm phase II clinical study to include 32 patients with advanced pancreatic cancer with KRAS G12D mutation to evaluate the effectiveness of HRS-4642 combined with nitutuzumab and AG for first-line treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study used a Simon two-stage design, with at least 15 subjects enrolled in the first stage. During this period, after 6-9 subjects complete the first cycle of treatment, the existing safety data shall be summarized and analyzed to integrate the safety results to assess the tolerance. If tolerated, the proposed dose, other dose level or dosage regimen shall be discussed by investigators. As with> 5 achieved remission (CR / PR), enrollment continued to 32; if 5 were remitted, the SMC assessed assessed and decided. The study process included screening, treatment and follow-up periods (safety and survival follow-up after termination of study treatment).

ELIGIBILITY:
Inclusion Criteria:

1.Age: 18-75 (including 18 and 75); 2.Metastatic pancreatic cancer (from pancreatic ductal epithelium); 3.Tumor tissue contains KRAS G12D mutation; 4.No systemic antitumor therapy in advanced stage; if previous neoadjuvant / adjuvant therapy, last treatment should be over 6 months; 5.At least one measurable lesion according to the RECIST v1.1 criteria; 6.The ECOG (Eastern Cooperative Oncology) score was 0-1; 7.Expected survival period of 3 months; 8.The functions of vital organs meets the following requirements (any blood components, cell growth factors are not allowed 2 weeks prior to enrollment):

1. Neutrophil count≥1.5×10^9 / L;
2. Platelet≥100×10^9 / L;
3. Hemoglobin≥100 g / L;
4. Serum albumin≥30 g / L;
5. Total bilirubin≤1.5×ULN; ALT, AST≤3×ULN and ALP≤2.5×ULN; if the patient has liver metastasis, ALT, ALT and AST≤5×ULN; if the patient has liver or bone metastasis, ALP≤5×ULN;
6. Creatinine clearance≥50 mL/min or serum creatinine ≤1.5×ULN;
7. Urinary protein <2+; if urine protein≥2+, an additional 24 hours urine protein quantification should be tested, and if 24 hours urine protein quantification <1g can be enrolled;
8. ECG: QTcF≤450 ms (male), QTcF≤470 ms (female);
9. Cardiac color ultrasound: LVEF (left ventricular ejection fraction) ≥50%; 9.Women of childbearing age must have a blood pregnancy test within 7 days before enrollment, the result should be negative and must be non-lactating and should be willing to use appropriate contraception during the trial and within 6 months of treatment. For men, surgical sterilization or consent to use appropriate contraception during the study and within 6 months after completion of treatment.

10.Volunteer to participate in the study and sign the informed consent form, good compliance, agreed to cooperate with the follow-up.

Exclusion Criteria:

1.Previous treatment:

1. Previous treatment of targeted therapy against KRAS G12D.
2. Previous targeted therapy against EGFR.
3. Received major surgery or major trauma within 4 weeks before enrollment, or palliative local treatment (including but not limited to palliative radiotherapy, interventional therapy) within 2 weeks prior to enrollment.
4. Have received any other clinical study medication within 4 weeks before enrollment, except for an observational (non-interventional) clinical study or interventional clinical study follow-up.

(5)14 days before enrollment with drugs that strongly inhibit or induce the hepatic drug-metabolizing enzymes CYP3A4 or CYP2C8.

2.The presence of a central nervous system (CNS) metastases. 3.Acute or chronic pancreatitis requiring clinical intervention. 4.Symptoms and signs of gastrointestinal obstruction or obstruction within 6 months before initiation of study treatment but can be screened if surgery is performed and the obstruction is completely resolved.

5.Within 2 weeks prior to enrollment, there is a third space effusion (such as a large amount of pleural fluid, ascites, etc.) that can not reach the stable state (no intervention treatment is needed after the removal of the drainage tube), and only a small amount of effusion on imaging and without clinical symptoms can be enrolled.

6.Severe infection occurred within 4 weeks before enrollment, such as severe pneumonia, bacteremia, infectious complications, requiring hospitalization; fever of unknown cause> 38.5℃ within 2 weeks before enrollment (fever caused by the tumor according to the investigator); 2 weeks of enrollment (except in cases of prophylactic antibiotics).

7.Severe cardiovascular and cerebrovascular disease. 8.Patients with known or suspected interstitial pneumonia except only interstitial changes on imaging.

9.Prior history of clear neurological or psychiatric disorders, including epilepsy and dementia.

10.Presence of non-healing wounds (severe, non-healing or split), uncured fractures.

11.Adverse events due to prior treatment prior to enrollment did not return to NCI-CTCAE level 1 (except for alopecia and enrollment criteria; except AEs not affecting the study medication).

12.Malignant tumors other than the primary tumor within the 5 years before enrollment, except those with low risk of metastasis and death: adequately treated cervical carcinoma in situ, skin basal cells or squamous cell carcinoma, etc.

13.Combined with active hepatitis B (hepatitis B surface antigen positive and HBV DNA 500 IU / mL), hepatitis C (hepatitis C antibody positive, and HCV-RNA above the lower limit of detection of the analytical method). Those known to have acquired immunodeficiency syndrome or test positive for HIV, and those infected with active syphilis. Subjects with active tuberculosis or a history of active tuberculosis infection within 48 weeks before screening, with or without treatment.

14.Known to be allergic to any component of HRS-4642; allergic to any component of nytuzumab or other monoclonal antibody / fusion proteins, albumin paclitaxel, gemcitabine.

15.By the investigator, the patient had other factors that might affect the study results or lead to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during the whole study

SECONDARY OUTCOMES:
Duration of remission （DoR） | Up to 2 years
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause during the whole study.
Disease control rate (DCR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during the whole study.
Progression-free survival （PFS） | Up to 2 years
  The time from enrolled to disease pregression or death from any cause during the whole study.
Overall survival (OS) | Up to 2 years
  The time from enrolled to death from any cause during the whole study.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang